CLINICAL TRIAL: NCT06236737
Title: Comparison of Sensorimotor and Yoga Exercise in Patients With Chronic Neck Pain
Brief Title: Sensorimotor Exercises and Neurodevelopmental Yoga in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Dilanur Özkaraoğlu, PT, MSc, PT,MSc, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MedipolU-FTR-DO-01
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Neck Pain
Keywords: Rehabilitation; Pain; Yoga; Proprioception
MeSH Terms: conditions — Neck Pain; Pain

STUDY DESIGN:
Intervention Model Description: Two intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensorimotor Exercise Group (Experimental): Sensorimotor exercise group; oculomotor exercise to provide information from the visual system, laser target exercise to provide information from the proprioception system, and postural stability exercise to provide information from the vestibular system. Within the scope of oculomotor exercise, gaze stability exercise and head-body coordination exercise will be given to the participants. Laser target exercise will be given with the laser target fixed on the participant's head and 90 cm away from the target. Postural stability exercise will be given in the form of tandem exercise and standing on one leg.
  Interventions: Other: Sensorimotor Exercise
- Yoga Exercise Group (Experimental): Yoga group will be given yoga exercises including 14 poses. These exercises are: bridge pose, corpse pose, bharadvaja's twist, downward facing dog, downward facing hero, extended side angle, extended triangle, mountain pose, prosperous pose, reclining big toe, standing half forward bend, thunderbolt pose, upward hand
  Interventions: Other: Yoga Exercise

INTERVENTIONS:
Other: Sensorimotor Exercise — The sensorimotor group was given oculomotor, gaze stability and postural stability exercises. Each session lasted 40 minutes in total.
  Arms: Sensorimotor Exercise Group
Other: Yoga Exercise — A flow was created for the yoga group. Each session lasting 40 minutes was included ocular motor, balance, meditation and stretching. Practices illustrated in table one were repeated for the eight weeks. Beginning of each session was focused on breathing exercises and the yoga flow is designed. Weeks 1-2. were prepared by focusing mostly on sagittal plane asanas. While 3-5. tweeks were focused on frontal plane asanas, 6-8. weeks were focused on transvers plan. Each session commenced with a 5-minute practice of a three dimensional breathing technique. This was followed by a 25-minute yoga asana flow, concluding with a 10-minute meditation in shavasana, also known as Corpse Pose. NDY was taught by an academician physiotherapist who has completed graduation in yoga therapy.
  Arms: Yoga Exercise Group

SUMMARY:
Neck pain is an important public health problem with a high lifetime prevalence and frequently occurring in all industrialized countries. Clinical practice guidelines for chronic neck pain recommend conservative management. Conservative treatment includes many approaches such as endurance, stretching and strengthening exercises, manual therapy, proprioceptive exercises, pilates and yoga. In patients with chronic neck pain, atrophy of deep neck muscles, deterioration in fiber type ratio, muscle tenderness and decreased range of motion are observed. These problems cause poor cervical postural control system and thus impaired sense of proprioception, loss of balance, decreased eye movement and cervical muscle activity. Sensorimotor control of upright posture and head-eye movement relies on information from the vestibular, visual, and proprioceptive systems that assemble throughout the central nervous system.The cervical spine has an important role in providing proprioceptive input. This role is associated with an abundance of cervical mechanoreceptors. Recent studies have shown that proprioceptive training is associated with cervical joint position sense, joint range of motion, pain and disability. Also yoga combines physical exercises with breathing techniques and meditation and yoga is one of the most commonly used complementary treatments for neck pain.The aim of study is to determine the effectiveness of exercises for sensorimotor structure and yoga exercises with physical and meditative effects in individuals with chronic neck pain.

DETAILED DESCRIPTION:
Participants diagnosed with chronic neck pain will be randomly divided into two groups as sensorimotor exercise group and yoga group by the evaluator. Sensorimotor exercise group; oculomotor exercise to provide information from the visual system, laser target exercise to provide information from the proprioception system, and postural stability exercise to provide information from the vestibular system. Yoga group will be given yoga exercises. Within the content of oculomotor exercise, gaze stability exercise and head-body coordination exercise will be given to the participants. Laser target exercise will be given with the laser target fixed on the participant's head and 90 cm away from the target. Postural stability exercise will be given in form of tandem exercise and standing on one leg. Yoga exercises will be applied by changing and combining 14 poses every week. The study will take 8 weeks. Participants in both groups will also be treated for 2 days a week. Participants will be evaluated twice, before and after treatment. Participants will be evaluated with Demographic Information Form, SF-36 Quality of Life Scale, Neck Disability Questionnaire, Tampa Kinesiophobia Scale, Numerical Pain Scale, Joint Range of Motion Measurement (G-Pro), Joint Position Error Test. Data analysis of the study will be done using SPSS 22.0 package program. The difference between Independent Groups will be compared with the Student's-t independent Test.

ELIGIBILITY:
Inclusion Criteria:

* aged 24-60 years of either sex, at least a 12 weeks history of CNP, CNP according to the Quebec Task Force grading system in Grade 1 and 2

Exclusion Criteria:

* according to Quebec Task Force grading system Grade 3 and 4 neck pain, neurological defects, speech and perception disorders, psychiatric diagnosis, recent history of neck trauma, recent history of cancer, diagnosed vestibular disorder, participants who diagnosed eye disorders, recent history of surgery, contraindications to yoga.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Cervical Joint Position Error Test | 8 weeks
  Cervical joint position error (JPE) test was used a laser pointer. A laser pointer was mounted onto a lightweight headband is then placed on the patient's head. The patient was sut 90 cm from the wall, and the started point (center of target or reference point) of the laser projection was marked. The participant (blindfolded or closed) performed active neck movement and then returned to the starting position as accurately as possible. The final laser position was measured relative to the starting position (distance or angle). The errors was measured after cervical extension, flexion, lateral flexions, and rotations.

SECONDARY OUTCOMES:
Range of Motion (ROM) | 8 weeks
  ROM was measured using the G-pro app installed on the iPhone 13. The examiner activated the G-pro app and pressed the "device axis" button to adjust the axis according to the test condition. For measuring flexion and extension, the iPhone was placed just beside the external auditory meatus and one axis of the app was aligned with the imaginary line between the base of the nostril and the external auditory meatus. Active lateral flexion ROM was measured in the sitting position. The center of the app was placed over the C7 spinous process, and one axis of the app was aligned with the occipital protuberance. Finally, because of difficulty in using the app for measuring active cervical rotation in sitting, this movement was evaluated in the supine position. The center of the app was positioned at the center of the head and one axis was aligned with the nose.
Numerical Pain Rating Scale (NPRS) | 8 weeks
  The 11-point numerical pain rating scale (NPRS) is a measure of pain in which participants rate their pain ranging from 0 (no pain) to 10 (worst imaginable pain),1-4 and it has been shown to have concurrent and predictive validity as a measure of pain intensity. The NPRS is as a valuable and dependable assessment tool that significantly complements comprehensive research and practices related to neck pain.
Neck Disability Index (NDI) | 8 weeks
  The NDI has 10 questions scored on a Likert scale (0 to 5), with higher total scores out of 50 indicating greater levels of perceived difficulty with activities of daily living due to neck pain. The NDI is a commonly used clinical outcome measure with good internal consistency and good construct validity
Tampa Scale for Kinesiophobia (TSK) | 8 weeks
  The TSK is a reliable and valid measurement tool that provides therapists valuable information on activity avoidance and pathological somatic focus in patients with musculoskeletal pain. It is a 17-questions scale calculated with Likert scoring and includes the parameters of re-injury and fear in work-related activities. The scoring is; "I strongly disagree" is 1, "I disagree" is 2, "I agree" is 3, "I strongly agree" is 4. A total score is calculated after reversing the fourth, eighth, twelfth and sixteenth items. A higher score on the scale indicates a higher level of kinesiophobia.
Quality of Life (Short Form-36) | 8 weeks
  The quality of life questionnaire (SF-36) was used to evaluate the patients' life quality with a mental and physical score. The SF-36 has been also used to test the correlation between health-related quality of life and related factors (sex, age, physical function, and daily functioning) rated on a 5-point scale. It consists of 36 items and 8 scales, including physical function, physical role, body pain, general health, vitality, social behavior, emotional role, and mental health. The obtained scores range between 0 and 100 with higher scores indicating better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Dilanur Kutlu Özkaraoğlu, MsC, Principal Investigator — Istanbul MedipolUniversity
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No